CLINICAL TRIAL: NCT06540079
Title: BIOTRONIK Conduction System Pacing With the Solia Lead
Brief Title: BIOTRONIK Conduction System Pacing With the Solia Lead - Solia CSP S
Acronym: BIO-CONDUCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G210349-Solia CSP S
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Sinus Node Dysfunction; Bradycardia; Atrioventricular Block
MeSH Terms: conditions — Sick Sinus Syndrome; Bradycardia; Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Solia CSP S LBB Lead (Experimental)
  Interventions: Device: Solia CSP S lead

INTERVENTIONS:
Device: Solia CSP S lead — The Solia CSP S pacing lead will be implanted in the LBBA for patients who meet all inclusion/exclusion criteria and give written informed consent.

SUMMARY:
The purpose of the BIO-CONDUCT study is to demonstrate the safety and effectiveness of the BIOTRONIK Solia CSP S pacing lead when implanted in the left bundle branch area (LBBA). Safety will be assessed by evaluating serious adverse device effects that occur through 3 months post-implant. Efficacy will be assessed by evaluating implant success rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for implantation of a BIOTRONIK pacemaker system, per standard guidelines. Single chamber, dual chamber, and CRT-P systems are allowed.
* Patient has an implant planned to utilize left bundle branch area (LBBA) pacing within 30 days of consent
* Patient is able to understand the nature of the study and provide written informed consent
* Patient is available for follow-up visits on a regular basis for the expected duration of follow-up
* Patient accepts Home Monitoring® concept
* Patient age is greater than or equal to 18 years at time of consent

Exclusion Criteria:

* Patient meets a standard contraindication for pacemaker system implant
* Patient is currently implanted with a pacemaker or ICD device
* Patient has had a previous unsuccessful attempt to place a lead in the LBBA
* Patient has planned cardiac surgical procedures or interventional measures within 3 months after implant
* Patient is expected to receive a heart transplant within 12 months
* Patient life expectancy less than 12 months
* Patient has the presence of another life-threatening, underlying illness separate from their cardiac disorder
* Patient reports pregnancy at the time of enrollment
* Patient is enrolled in any other investigational cardiac clinical study during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Device Effect (SADE)-Free Rate at 3 Months | 3 months post-implant
  Serious adverse device effect includes both serious lead related and serious implant related device effects. The overall percentage of subjects without serious lead related adverse device effects related to Solia CSP S lead utilized or attempted to be implanted in the LBBA and serious implant procedure events related to the Solia CSP S LBBA lead will be reported.
Implant Success Rate | At implant procedure
  The overall percentage of subjects with successful placement of Solia CSP S lead in LBBA will be reported.

SECONDARY OUTCOMES:
Quality of Life (QOL) from Baseline through 12 Months Post-Implant | 12 months post-implant
  This secondary outcome will evaluate the improvement in QOL for subjects with the Solia CSP S lead implanted in the LBBA. The parameter of interest is the change in the physical function SF-36 (36-Item Short Form Health Survey) QOL scale from pre-implant baseline to 12 months post-implant, which will be calculated as the mean change from baseline for all subjects that complete both the baseline QOL and 12-month QOL questionnaire. Note that all items are scored so that a high score defines a more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Serious Adverse Device Effect (SADE)-Free Rate at 6 Months | 6 months post-implant
  Serious adverse device effect includes both serious lead related and serious implant related device effects. The overall percentage of subjects without serious lead related adverse device effects related to Solia CSP S lead utilized or attempted to be implanted in the LBBA and serious implant procedure events related to the Solia CSP S LBBA lead will be reported.
Serious Adverse Device Effect (SADE)-Free Rate at 12 Months | 12 months post-implant
  Serious adverse device effect includes both serious lead related and serious implant related device effects. The overall percentage of subjects without serious lead related adverse device effects related to Solia CSP S lead utilized or attempted to be implanted in the LBBA and serious implant procedure events related to the Solia CSP S LBBA lead will be reported.
Pacing Threshold Measurements at 3 Months | 3 months post-implant
  Pacing threshold measurements for Solia CSP S leads implanted in the LBBA at the 3 month follow-up visit.
Sensing Measurements at 3 Months | 3 months post-implant
  R-wave sensing amplitude measurements for Solia CSP S leads implanted in the LBBA at the 3 month follow-up visit.
Pacing Impedance at 3 Months | 3 months post-implant
  Pacing impedance measurements for Solia CSP S leads implanted in the LBBA at the 3 month follow-up visit.
Pacing Threshold Measurements at 6 Months | 6 months post-implant
  Pacing threshold measurements for Solia CSP S leads implanted in the LBBA at the 6 month follow-up visit.
Sensing Measurements at 6 Months | 6 months post-implant
  R-wave sensing amplitude measurements for Solia CSP S leads implanted in the LBBA at the 6 month follow-up visit.
Pacing Impedance at 6 Months | 6 months post-implant
  Pacing impedance measurements for Solia CSP S leads implanted in the LBBA at the 6 month follow-up visit.
Pacing Threshold Measurements at 12 Months | 12 months post-implant
  Pacing threshold measurements for Solia CSP S leads implanted in the LBBA at the 12 month follow-up visit.
Sensing Measurements at 12 Months | 12 months post-implant
  R-wave sensing amplitude measurements for Solia CSP S leads implanted in the LBBA at the 12 month follow-up visit.
Pacing Impedance at 12 Months | 12 months post-implant
  Pacing impedance measurements for Solia CSP S leads implanted in the LBBA at the 12 month follow-up visit.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Banner - University Medical Center Phoenix, Phoenix, Arizona
  - Cardiology Associates Medical Group, Ventura, California
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - NYU Heart Rhythm Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Atrium Health Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cardiology Consultants of Philadelphia, Paoli, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant level data collected within the study will be shared for approved requests.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available beginning no later than 12 months and ending 3 years after study completion.
Access Criteria: Proposals should be directed to BIOTRONIK Clinical Studies (BIOTRONIK Inc., Attn: Clinical Studies, 6024 Jean Road, Lake Oswego, OR; 1-800-547-0394). BIOTRONIK, in consultation with the National Principal Investigator, will review and critique requests for scientific merit, fiscal feasibility, and logistical feasibility. If approved, the data requestors will need to sign a data use/access agreement prior to obtaining the data. BIOTRONIK reserves the right to delete any confidential information or other proprietary information (including trade secrets and patent protected materials) from the shared information.